CLINICAL TRIAL: NCT04926337
Title: Preoxygenation With High-flow Nasal Oxygen in Comparison to Standard Face Mask in Adult Trauma Patients During Rapid Sequence Induction Anesthesia- a Prospective, Non-randomized, Before-and-after Study
Brief Title: Preoxygenation With High-flow Nasal Oxygen in Adult Trauma Patients During Rapid Sequence Induction Anaesthesia
Acronym: PRIOR-Trauma
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Senior consultant, Associate Professor, Karolinska University Hospital
Other Study IDs: PRIOR-Trauma
Record Dates: First submitted 2021-06-07; First posted 2021-06-15 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia; Hypoxia; Trauma; Rapid Sequence Induction
MeSH Terms: conditions — Hypoxia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tight fitting facemask: Preoxygenation with tight facemask, 100% oxygen.
  Interventions: Device: Tight Fitting Facemask
- High flow nasal oxygen: Preoxygenation with high flow nasal oxygen, 100% oxygen
  Interventions: Device: High Flow Nasal Oxygen (HFNO)

INTERVENTIONS:
Device: Tight Fitting Facemask — Preoxygenation with tight facemask, 10 L/min, 100% oxygen.
  Groups: Tight fitting facemask
Device: High Flow Nasal Oxygen (HFNO) — Preoxygenation with high flow nasal oxygen, 40-70 L/min, 100% oxygen.
  Groups: High flow nasal oxygen

SUMMARY:
Previous studies investigating apnoea oxygenation has shown that delivering oxygen via a high flow can maintain adequate oxygen saturation levels in a patient for over 30 minutes.

It has recently been demonstrated, in several studies, that High Flow Nasal Oxygen (HFNO) used during preoxygenation in patients undergoing emergency surgery is at least equally effective as preoxygenation with standard tight fitting mask. Data from these recent studies investigating arterial oxygen saturation levels during rapid sequence induction anaesthesia have not been able to detect any difference between the two methods. The mean apnea time among the patients in the previous studies have been relatively short.

Patients suffering traumatic injuries could be more prone to desaturate during prolonged apnea due to being hemodynamic unstable or suffering injuries to the respiratory tract.

Based on the above, the aim is now to conduct a trial where trauma patients are preoxygenated with high flow nasal oxygen before anaesthetised with rapid sequence induction (RSI) technique. The trial is set to be a before-and-after study. During approximately 6 to 9 months data will be registered from trauma patients undergoing emergency anaesthesia where preoxygenation is performed according to standard rutin, with traditional facemask. During the coming six to nine months trauma patients undergoing emergency anaesthesia will be preoxygenated with high flow nasal oxygen. Data will be registered and compared to the data collected from the patients preoxygenated with facemark.

The general purpose of this project is to compare the preoxygenation technique based on HFNO with traditional preoxygenation with a tight fitting mask, with the main focus being oxygen saturation levels, during rapid sequence induction (RSI) intubation in trauma patients in need of immediate anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 1 Adult, ≥18 years old
* 2 Level 1 trauma with patients in need of emergency anaesthesia before leaving the trauma unit (trauma room or nearby operating theatre).

Exclusion Criteria:

* 1 Patients with or with risk of skull or facial injuries where application of nasal cannula is decided to be avoided by the trauma team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligable patients suffering Level 1 trauma and in need of emergency anaesthesia will be included.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with a peripheral oxygen saturation (SpO2) below 93% | From start of anaesthesia until 1 minute after tracheal intubation.
  Compare the number of patients with a peripheral oxygen saturation (SpO2) below 93% from induction of anesthesia (when induction drug is administered) until one minute after intubation between the group preoxygenated using HFNO and the group preoxygenated with traditional tight-fitting mask.

SECONDARY OUTCOMES:
Lowest median SpO2. | From start of anaesthesia until 1 minute after tracheal intubation.
  Lowest median SpO2 during preoxygenation using HFNO compared to traditional preoxygenation from when first anesthetic drug is administered until 1 minute after intubation
End tidal gas levels | At the first breath after tracheal intubation.
  Difference in levels of ETO2 and ETCO2 in the first breath after intubation with HFNO oxygenation compared to traditional pre-oxygenation.
Time span from start of preoxygenation until intubation. | Could vary depending on patient and trauma, from a couple of minutes up to 20-30 minutes.
  Compare the time span from start of preoxygenation until intubation between the HFNO group and the group with traditional preoxygenation.
Time span from entering trauma room until intubation. | Could vary depending on patient and trauma, from a couple of minutes up to an hour.
  Time span from when the patient enters the trauma room until intubation in the HFNO group compared to the group with traditional preoxygenation.
Difficulties with induction of anaesthesia | Could vary depending on patient and trauma, from a couple of minutes up to 20-30 minutes.
  Compare the perceived difficulties during induction of anaesthesia between the HFNO technique and traditional preoxygenation, for example tolerance to mask or nasal cannula
Frequency of complications | Could vary depending on patient and trauma, from a couple of minutes up to 20-30 minutes.
  Frequency of complications (aspiration, signs of intraabdominal/intracranial gas, difficulties intubating the trachea, hypotension) in the HFNO group compared to the group preoxygenated with traditional facemask.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided